CLINICAL TRIAL: NCT02230865
Title: Prediction of Acute Postoperative Pain and Analgesic Consumption by Preoperative Responses to Experimental Pain in Patients Undergoing Chest Wall Surgery
Brief Title: Prediction of Acute Postoperative Pain and Analgesic Consumption
Acronym: MIRPEX-3
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kasper Grosen (Other)
Responsible Party: Sponsor-Investigator, Kasper Grosen, PhD, Aarhus University Hospital
Organization: University of Aarhus (Other)
Other Study IDs: MIRPEX-3
Record Dates: First submitted 2014-08-29; First posted 2014-09-03 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Postoperative Pain
Keywords: Funnel chest (Pectus excavatum)
MeSH Terms: conditions — Pain, Postoperative; Funnel Chest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgery: Minimally invasive repair of pectus excavatum

SUMMARY:
Pain is an expected part of surgical recovery but effective pain management remains challenging. The high variability in postoperative pain experience and analgesic treatment response between patients is part of the challenge. Few studies have yet combined preoperative assessment of responses to experimental pain with measurements of cognitive and emotional processes in the prediction of postoperative pain.

We hypothesize, that preoperative evoked brain potentials (using standard electroencephalographic brain imaging), endogenous pain inhibition capacity (conditioned pain modulation), responses to pressure/thermal pain stimulation, and/or situational pain-related catastrophic thinking are useful clinical predictors of postoperative pain and analgesic consumption.

DETAILED DESCRIPTION:
Preselected preoperative predictor variables/individual patient characteristics include the following:

* Evoked brain potentials (using standard electroencephalographic brain imaging)
* Capacity of descending pain inhibition induced by a cold pressor test (2C in 120 sec)
* Pressure pain detection and tolerance thresholds in muscle (m.quadriceps)
* Pressure pain tolerance thresholds in bone (sternum and tibia)
* Heat pain tolerance threshold in skin (forearm)
* Responses to the Situational and Dispositional Pain Catastrophizing Scale
* Response to the State-Trait and Anxiety Inventory
* Response to the Beck's Depression Inventory

ELIGIBILITY:
Inclusion Criteria:

* Elective minimally invasive surgical correction of funnel chest (pectus excavatum
* age ≥15 years.

Exclusion Criteria:

* Previous thoracic surgical interventions
* Presence of diseases affecting the central and/or peripheral nervous system
* Presence of chronic pain conditions
* Inability to speak and/or understand Danish
* Inability to understand and participate in the experimental pain session
* Presence of psychiatric disorders
* History of frostbite in the non-dominant upper limb
* Presence of sores or cuts on non-dominant upper limb
* Presence of cardiovascular disease
* History of fainting and/or seizures
* Presence of fractures of the non-dominant upper limb
* Presence of Reynaud's phenomenon.

Secondary exclusions included:

* Insensitivity to experimental cold pressor pain
* Lack of epidural catheter placement
* Re-operation

Min Age: 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with funnel chest (pectus excavatum) undergoing corrective chest wall surgery at Aarhus University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain intensity | Within the first 5 days after surgery
  11-point (0-10) numerical rating scale of pain intensity
Postoperative pain unpleasantness | Within the first 5 days after surgery
  11-point (0-10) numerical rating scale of pain unpleasantness
Postoperative consumption of analgesics | Within the first 5 days after surgery
  The use of all pain-related treatments, including rescue analgesics and any other concomitant pain treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Asbjørn M Drewes, MD, PhD, DMSci, Study Director — Mech-Sense, Department of Gastroenterology, Aalborg University Hospital, Denmark; Kasper Grosen, MHSc, PhD, Principal Investigator — Department of Cardiothoracic and Vascular Surgery, Aarhus University Hospital, Denmark; Hans K Pilegaard, MD, Study Chair — Department of Cardiothoracic and Vascular Surgery, Aarhus University Hospital, Denmark; Lene Vase, MSc (Psychology), PhD, Study Chair — Department of Psychology, Aarhus University, Denmark; Mogens Pfeiffer-Jensen, MD, PhD, Study Chair — Aarhus University Hospital; Vibeke E Hjortdal, MD, PhD, DMSci, Study Chair — Department of Cardiothoracic and Vascular Surgery, Aarhus University Hospital, Denmark; Anne E Olesen, PhD, Study Chair — Mech-Sense, Department of Gastroenterology, Aalborg University Hospital, Denmark; Mikkel Gram, MScEE, Study Chair — Mech-Sense, Department of Gastroenterology, Aalborg University Hospital, Denmark
Locations (1):
- Deparment of Cardiothoracic and Vascular Surgery, Aarhus University Hospital, Denmark, Aarhus, Denmark

REFERENCES:
- [Background] Grosen K, Vase L, Pilegaard HK, Pfeiffer-Jensen M, Drewes AM. Conditioned pain modulation and situational pain catastrophizing as preoperative predictors of pain following chest wall surgery: a prospective observational cohort study. PLoS One. 2014 Feb 26;9(2):e90185. doi: 10.1371/journal.pone.0090185. eCollection 2014. PMID 24587268
- See also: Related Info — http://www.mech-sense.com